CLINICAL TRIAL: NCT07317908
Title: Effects of 10 Weeks of Zumba Training on Anxiety and Depression: A Randomized Controlled Trial
Brief Title: Effects of a 10-Week Zumba Program on Anxiety and Depression in Adults
Acronym: ZUMBA-AN-DE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manuel Jesús Rodríguez Chavarría (Other)
Responsible Party: Sponsor-Investigator, Manuel Jesús Rodríguez Chavarría, Principal Investigator, Universidad de Extremadura
Organization: Universidad de Extremadura (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZU-AN-DE
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Anxiety; Depression; Psychological Well-being
Keywords: zumba; Physical exercise; Aerobic exercise; mental health; Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression; Psychological Well-Being; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants were randomly allocated to one of two parallel groups: a Zumba intervention group or a control group. The intervention group participated in supervised Zumba sessions three times per week for 10 weeks, while the control group maintained their usual lifestyle without structured exercise.
Masking Description: This was an open-label study. Due to the nature of the exercise intervention, neither participants nor investigators were blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zumba Group (Experimental): Participants assigned to the experimental group formed the Zumba intervention group. This group followed a supervised Zumba-based exercise program over a period of 10 weeks. The intervention consisted of structured group sessions performed several times per week and led by a qualified instructor. Sessions were based on choreographed aerobic dance movements performed to music, providing moderate-to-vigorous intensity physical activity aimed at improving cardiovascular fitness and overall physical engagement.
  Interventions: Behavioral: Zumba-based Exercise Program
- Group Control (No Intervention): Participants in the control group did not participate in the exercise intervention and were instructed to maintain their usual lifestyle and physical activity habits throughout the study period.

INTERVENTIONS:
Behavioral: Zumba-based Exercise Program — Participants assigned to this intervention received a supervised Zumba-based exercise program lasting 10 consecutive weeks. The intervention consisted of group-based aerobic dance sessions conducted several times per week and led by a qualified instructor. Sessions included choreographed dance movements performed to music, designed to elicit moderate-to-vigorous physical activity and to promote cardiovascular fitness and overall physical engagement. The program followed a standardized structure across sessions and was implemented as the sole intervention during the study period.
  Arms: Zumba Group

SUMMARY:
This randomized controlled trial aimed to examine the effects of a 10-week Zumba exercise program on anxiety and depression levels in healthy adults. Participants aged 40 to 65 years were randomly assigned to either a Zumba intervention group or a control group that maintained their usual lifestyle. The intervention consisted of three supervised Zumba sessions per week, each lasting approximately 50 minutes. Anxiety and depression were assessed before and after the intervention using the Hospital Anxiety and Depression Scale (HADS). The study sought to determine whether a structured, group-based aerobic exercise program could improve psychological well-being in a non-clinical adult population.

DETAILED DESCRIPTION:
This study was designed as a randomized controlled trial to investigate the impact of a structured Zumba exercise program on anxiety and depression in healthy adults. Participants were recruited from the community and randomly allocated to either a Zumba intervention group or a control group.

The intervention group participated in a 10-week Zumba program, consisting of three supervised sessions per week. Each session lasted approximately 50 minutes and was conducted at moderate intensity, monitored using the Borg Rating of Perceived Exertion scale. Sessions included a standardized warm-up, choreographed aerobic dance routines, and a cool-down period.

The control group was instructed to maintain their usual lifestyle and not to engage in any new structured exercise programs during the study period.

Anxiety and depression were assessed at baseline and after the intervention using the Hospital Anxiety and Depression Scale (HADS). All assessments were conducted under standardized conditions by trained researchers. The primary objective was to evaluate changes in anxiety and depression symptoms between groups following the intervention.

The study was conducted in accordance with ethical standards, and all participants provided written informed consent prior to participation.

ELIGIBILITY:
Inclusion Criteria:

* adults aged between 40 and 65 years
* not having regularly practised Zumba or other dance disciplines during the previous 12 months
* medical authorisation or absence of pathologies to participate in supervised physical activity

Exclusion Criteria:

* presence of orthopaedic, neurological, cardiorespiratory conditions or lack of standing stability that would prevent safe completion of the programme
* participation in any other structured exercise programme during the intervention period
* missing more than 10% of the total sessions (missing more than 2 sessions)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Anxiety and Depression | Baseline and Week 10 (end of intervention)
  Anxiety and depression were assessed using the Hospital Anxiety and Depression Scale (HADS), a validated self-report questionnaire designed to detect clinically relevant symptoms of anxiety and depression in non-psychiatric populations. The scale consists of 14 items divided into two subscales: anxiety (HADS-A) and depression (HADS-D), each ranging from 0 to 21 points, with higher scores indicating greater symptom severity. Total HADS scores range from 0 to 42. Changes in total and subscale scores were used to evaluate the effects of the intervention on psychological well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Osuna fitness, Osuna, Sevilla, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly. The dataset contains sensitive health-related information collected in a supervised exercise intervention and was obtained under informed consent that did not include data sharing. Data may be available from the corresponding author upon reasonable request, subject to ethical approval.